CLINICAL TRIAL: NCT06357091
Title: ACL Reconstruction With Human Allograft Cortical Bone Screw (Shark Screw®) or Biocomposite-interference Screws - a Prospective, Randomized, Controlled Trial.
Brief Title: ACL Reconstruction With Shark Screw® or Biocomposite-interference Screws
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Rofner-Moretti (Other)
Responsible Party: Sponsor-Investigator, Alexander Rofner-Moretti, Senior Physician Dr. med. Alexander Rofner-Moretti, Bezirkskrankenhaus Schwaz
Organization: Bezirkskrankenhaus Schwaz (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1097/2023 ACL-Shark Screw®
Record Dates: First submitted 2024-02-13; First posted 2024-04-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Reconstruction; Anterior Cruciate Ligament Injury
Keywords: ACL; tunnel widening; human allogeneic cortical bone screw; Shark Screw®; biotenodese screw; re-rupture rate; IKDC; KOOS; Lysholm Knee Score; Tegner Activity Score; range of motion (ROM)
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL reconstruction with human allogeneic cortical bone screw (Shark Screw®) (Experimental): The sugery techniqueis the same for both arms. An allograft screw (Shark Screw ACL®; Surgebright GmbH, A-4040 Lichtenberg, Austria) is used. At the beginning of the operation, the diagnosis is confirmed arthroscopically. The tendon is prepared. The bone tunnels will be created due to the size of the graft. The graft is pulled in and fixed with the intereference screw (Shark Screw ACL®). The tibial bone tunnel will be filled with cancellous chips. Finally, the graft is checked for strength and possible anterior or lateral pinching. The arthroscopic fluid is aspirated and the wound is closed.
  Interventions: Procedure: ACL reconstruction with Shark Screw ACL®
- ACL reconstruction with Mecta Composite interference screw (Active Comparator): The sugery techniqueis the same for both arms. A Mecta-composite-screw, (Medacta, Castello San Pietro, Swiss) is used. At the beginning of the operation, the diagnosis is confirmed arthroscopically. The tendon is prepared. The bone tunnels will be created due to the size of the graft. The graft is pulled in and fixed with the intereference screw (Mecta-composite-screw, Medacta). The tibial bone tunnel will be filled with cancellous chips. Finally, the graft is checked for strength and possible anterior or lateral pinching. The arthroscopic fluid is aspirated and the wound is closed.
  Interventions: Procedure: ACL reconstruction with biocomposite screw (Mecta)

INTERVENTIONS:
Procedure: ACL reconstruction with Shark Screw ACL® — ACL reconstruction with the Shark Screw ACL®, Investigation of tunnel widening
  Arms: ACL reconstruction with human allogeneic cortical bone screw (Shark Screw®)
Procedure: ACL reconstruction with biocomposite screw (Mecta) — ACL reconstruction with biocomposite screw (Mecta), Investigation of tunnel widening
  Arms: ACL reconstruction with Mecta Composite interference screw

SUMMARY:
The goal of this clinical trial is to compare the outcome of 2 different screws for Anterior cruciate ligament reconstruction. The main question is if the human allogeneic cortical bone screw reduces tunnel widening in comparison to conventional treatment with a biocomposite screw. Additional the re-rupture rate will be evaluated and knee scores will be recorded before surgery and after surgery. Participants will have MRI before and after surgery, 3, 6, 12, and 24 months after surgery and Computertomography after surgery, 3, 6 and 24 months after surgery. Questionnaires (Knee-scores) will be recorded before surgery, 6, 12, 24 months after surgery.

the investigators hope that with the human cortical bone screw the tunnel widening is reduced and the re-rupture rate is low

DETAILED DESCRIPTION:
Rupture of the anterior cruciate ligament of the knee joint is a common (sports) injury in young adults . Depending on various patient-related factors, such an injury can be treated surgically or conservatively . Arthroscopic and anatomical reconstruction is currently considered the gold standard of surgical treatment. In this procedure, the torn anterior cruciate tendon will be replaced usually with the own semitendinosus ligament, the patellar ligament or the quadriceps tendon by inserting it through bone tunnels in the femur and tibia.

However, the optimal technique for fixing the graft remains unclear. Until the replacement graft has healed, the suspension of the graft remains the weak point of the overall construct . The currently common procedures are fixation by means of interference screw in the bone tunnels and distal fixation using endobuttons. These fixation methods differ only insignificantly in clinical scores, stability, or failure rate .

A frequent complication after reconstruction of the anterior cruciate ligament is secondary tunnel dilatation, which has been described in up to 84% of cases. The cause of this is not yet fully understood. Nakazato et al. cites a longer graft and an increased dorsolateral tibial slope. Taketomi makes the posterior tibial slope particularly responsible for tibial tunnel widening and describes that an osteolysis process occurs due to the penetration of synovial fluid into the space between the tendon and the tunnel . Moon et al. see a negative correlation between the length of the graft insertion and tunnel dilation. The widening of the bone tunnels seem not to induce instability, but complicates a follow-up operation, e.g. a new cruciate ligament plasty in the event of rerupture following new trauma. The often up to twice as large bone tunnels make it difficult to find sufficient bone tissue to create a new tunnel. If the already existing and enlarged tunnel is reused, there is a risk of inadequate fixation and lack of incorporation of the new graft. In the revision, a two-stage procedure is often necessary, especially in the case of pronounced widening of the bone tunnel. The group postulates that with a tunnel width &gt;14 mm, only a two-stage procedure is possible. In a first operation, the bone tunnel must be filled with autologous or similar, and only in a second session a new reconstruction of the anterior cruciate ligament can be attempted.

the investigators are planning a prospective, randomized, controlled, single-blind and monocentric study with 2 parallel groups to investigate an alternative fixation method in cruciate ligament surgery. This involves a screw made from allogenic bone (Shark Screw ACL®; Surgebright GmbH, A-4040 Lichtenberg, Austria) in the form of an interference screw obtained from donor cortical bone. The insertion of this bone screw is identical to the usual interference screws. This type of osteosynthesis material has already proven in other forms in fracture treatment. The investigators have been using screws made from allogenic bone in a similar form for the treatment of scaphoid fractures for more than 4 years , Calcaneal fractures, corrective osteotomies, and arthrodesis with excellent success in everyday clinical practice. Treatment with an allogenic bone screw is compared with the current standard treatment with resorbable interference screw MectaScrew (composite), Medacta Int. Str. Regina 34, 6874 Castel San Pietro, Switzerland) in a control group. The aim is to include 80 patients who will be included in the study, i.e. 40 per group. Surgical method, treatment plan and follow up treatment do not differ.

The main objective of the planned study is to analyze the dilation of the bone tunnels in the two groups. This will be done by means of magnetic resonance imaging (MRI) and computer tomography (CT) examinations (MRI preoperatively, postoperatively (within 3 days) and at 6, 12 and 24 months after surgery, CT postoperatively within 3 days and at 6 and 24 months after surgery). The bone tunnels are measured and the results of the two groups are compared to determine whether the allograft screw shows less bone tunnel dilation than the current standard treatment. An initial evaluation of the data and publication is planned after 12 months; the final evaluation and publication will take place after 24 months. The secondary objectives are to record the advantages and disadvantages of the allografts and to analyze their safety and effectiveness. In particular, the incorporation of the screws is to be assessed and classified. In order to better assess the outcome of the operation, clinical parameters will be recorded, and the two groups compared with each other. Furthermore, MRI will be analyzed for its informative value with regard to bone tunnel measurement.

The null hypothesis is that the two surgical procedures (bone screw / biocomposite screw) do not differ in outcome. The alternative hypothesis is that the use of the human, allogenic cortical bone screw as a fixation element for anterior cruciate ligament reconstruction results in faster and, above all, better incorporation of the graft, with less widening of the bone tunnel. Based on the experience of the investigators with similar osteosynthesis material made from allogenic bone, it is to be expected that the bone tunnel will heal scare free. The investigators see the advantage of the proposed treatment particularly in its bone-sparing nature. It is to be expected that this will make possible revision easier and that a two-stage procedure will be necessary less often.

ELIGIBILITY:
Inclusion Criteria:

* MRI-verified rupture of the anterior cruciate ligament
* Indication for replacement surgery
* Surgery within 6 months of injury
* Uninjured contralateral knee

Exclusion Criteria:

* Previous rupture of the anterior cruciate ligament on the side to be operated on (rerupture)
* Primary bone disease
* inflammatory disease
* Unstable meniscus
* complete rupture of a collateral ligament
* early rerupture during the examination period (early rerupture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2034-01-31 (Estimated); Study Completion 2034-01-31 (Estimated)

PRIMARY OUTCOMES:
bone tunnel widening will be measured by CT and/or MRI and measured in mm | immadiately after surgery, 3, 6, 12 and 24 months after surgery.
  bone tunnel widening will be evaluated and measured by CT and/or MRI and measured in mm

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Scores | before surgery and 6, 12 and 24 months after surgery
  IKDC will be evaluated by questionnaires, it can be between 0 and 100 the higher the better is the outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) Scores | before surgery and 6, 12 and 24 months after surgery
  KOOS Score will be evaluated by questionnaires, it can be between 0 and 100 the higher the better is the outcome
Lysholm Knee Score | before surgery and 6, 12 and 24 months after surgery
  Lysholm Knee Score will be evaluated by questionnaires, one of the most frequently used assessment tools for the results of Anterior cruciate ligament reconstruction even though it only measures activities of daily living, it can be between 0 and 100 the higher the better is the outcome.
Tegner Activity Score | before surgery and 6, 12 and 24 months after surgery
  Tegner Activity Score will be evaluated by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rofner-Moretti, MD, Principal Investigator — Bezirkskrankenhaus Schwaz Betriebsgesellschaft m.b.H
Locations (1):
- Bezirkskrankenhaus Schwaz Betriebsgesellschaft m.b.H, Schwaz, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
due to sensitivity of individual data and data protection restrictions in Austria

REFERENCES:
- [Background] Hanslik-Schnabel B, Flory D, Borchert GH, Schanda JE. Clinical and Radiologic Outcome of First Metatarsophalangeal Joint Arthrodesis Using a Human Allogeneic Cortical Bone Screw. Foot Ankle Orthop. 2022 Jul 29;7(3):24730114221112944. doi: 10.1177/24730114221112944. eCollection 2022 Jul. PMID 35924004
- [Background] Krasny C, Radda C, Polke R, Schallmayer D, Borchert GH, Albrecht C. A human, allogeneic cortical bone screw for distal interphalangeal joint (DIP) arthrodesis: a retrospective cohort study with at least 10 months follow-up. Arch Orthop Trauma Surg. 2023 Jul;143(7):4557-4564. doi: 10.1007/s00402-023-04785-2. Epub 2023 Feb 9. PMID 36757467
- [Background] Sailer S, Lechner S, Flossmann A, Wanzel M, Habeler K, Krasny C, Borchert GH. Treatment of scaphoid fractures and pseudarthroses with the human allogeneic cortical bone screw. A multicentric retrospective study. J Orthop Traumatol. 2023 Feb 10;24(1):6. doi: 10.1186/s10195-023-00686-7. PMID 36765020
- [Background] Pastl K, Schimetta W. The application of an allogeneic bone screw for osteosynthesis in hand and foot surgery: a case series. Arch Orthop Trauma Surg. 2022 Oct;142(10):2567-2575. doi: 10.1007/s00402-021-03880-6. Epub 2021 Apr 8. PMID 33834287
- [Background] Brcic I, Pastl K, Plank H, Igrec J, Schanda JE, Pastl E, Werner M. Incorporation of an Allogenic Cortical Bone Graft Following Arthrodesis of the First Metatarsophalangeal Joint in a Patient with Hallux Rigidus. Life (Basel). 2021 May 24;11(6):473. doi: 10.3390/life11060473. PMID 34073841
- [Background] Pastl K, Pastl E, Flory D, Borchert GH, Chraim M. Arthrodesis and Defect Bridging of the Upper Ankle Joint with Allograft Bone Chips and Allograft Cortical Bone Screws (Shark Screw(R)) after Removal of the Salto-Prosthesis in a Multimorbidity Patient: A Case Report. Life (Basel). 2022 Jul 11;12(7):1028. doi: 10.3390/life12071028. PMID 35888116
- [Background] Mayr R, Smekal V, Koidl C, Coppola C, Eichinger M, Rudisch A, Kranewitter C, Attal R. ACL reconstruction with adjustable-length loop cortical button fixation results in less tibial tunnel widening compared with interference screw fixation. Knee Surg Sports Traumatol Arthrosc. 2020 Apr;28(4):1036-1044. doi: 10.1007/s00167-019-05642-9. Epub 2019 Aug 1. PMID 31372680
- [Background] Yumashev AV, Baltina TV, Babaskin DV. Outcomes after arthroscopic revision surgery for anterior cruciate ligament injuries. Acta Orthop. 2021 Aug;92(4):443-447. doi: 10.1080/17453674.2021.1897744. Epub 2021 Mar 19. PMID 33739222
- [Background] Webster KE, Feller JA, Hameister KA. Bone tunnel enlargement following anterior cruciate ligament reconstruction: a randomised comparison of hamstring and patellar tendon grafts with 2-year follow-up. Knee Surg Sports Traumatol Arthrosc. 2001;9(2):86-91. doi: 10.1007/s001670100191. PMID 11354858
- [Background] Linn RM, Fischer DA, Smith JP, Burstein DB, Quick DC. Achilles tendon allograft reconstruction of the anterior cruciate ligament-deficient knee. Am J Sports Med. 1993 Nov-Dec;21(6):825-31. doi: 10.1177/036354659302100611. PMID 8291633
- [Background] Fahey M, Indelicato PA. Bone tunnel enlargement after anterior cruciate ligament replacement. Am J Sports Med. 1994 May-Jun;22(3):410-4. doi: 10.1177/036354659402200318. PMID 8037283
- [Background] Taketomi S, Inui H, Yamagami R, Nakazato K, Kawaguchi K, Kono K, Sameshima S, Kage T, Tanaka S. Lateral posterior tibial slope does not affect femoral but does affect tibial tunnel widening following anatomic anterior cruciate ligament reconstruction using a Bone-Patellar Tendon-Bone graft. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2022 Oct 5;30:25-31. doi: 10.1016/j.asmart.2022.09.003. eCollection 2022 Oct. PMID 36254269
- [Background] Fauno P, Kaalund S. Tunnel widening after hamstring anterior cruciate ligament reconstruction is influenced by the type of graft fixation used: a prospective randomized study. Arthroscopy. 2005 Nov;21(11):1337-41. doi: 10.1016/j.arthro.2005.08.023. PMID 16325084
- [Background] Lee DK, Kim JH, Lee BH, Kim H, Jang MJ, Lee SS, Wang JH. Influence of Graft Bending Angle on Femoral Tunnel Widening After Double-Bundle ACL Reconstruction: Comparison of Transportal and Outside-In Techniques. Orthop J Sports Med. 2021 Oct 22;9(10):23259671211035780. doi: 10.1177/23259671211035780. eCollection 2021 Oct. PMID 34708137
- [Background] Moon HS, Choi CH, Yoo JH, Jung M, Lee TH, Choi KH, Kim SH. The Graft Insertion Length in the Femoral Tunnel During Anterior Cruciate Ligament Reconstruction With Suspensory Fixation and Tibialis Anterior Allograft Does Not Affect Surgical Outcomes but Is Negatively Correlated With Tunnel Widening. Arthroscopy. 2021 Sep;37(9):2903-2914.e1. doi: 10.1016/j.arthro.2021.03.072. Epub 2021 Apr 20. PMID 33887417
- [Background] Nakazato K, Taketomi S, Inui H, Yamagami R, Kawaguchi K, Tanaka S. Lateral posterior tibial slope and length of the tendon within the tibial tunnel are independent factors to predict tibial tunnel widening following anatomic anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2021 Nov;29(11):3818-3824. doi: 10.1007/s00167-020-06419-1. Epub 2021 Jan 18. PMID 33459832
- [Background] Cavaignac E, Mesnier T, Marot V, Fernandez A, Faruch M, Berard E, Sonnery-Cottet B. Effect of Lateral Extra-articular Tenodesis on Anterior Cruciate Ligament Graft Incorporation. Orthop J Sports Med. 2020 Nov 30;8(11):2325967120960097. doi: 10.1177/2325967120960097. eCollection 2020 Nov. PMID 33299900
- [Background] de Beus A, Koch JE, Hirschmann A, Hirschmann MT. How to evaluate bone tunnel widening after ACL reconstruction - a critical review. Muscles Ligaments Tendons J. 2017 Sep 18;7(2):230-239. doi: 10.11138/mltj/2017.7.2.230. eCollection 2017 Apr-Jun. PMID 29264333
- [Background] Han DL, Nyland J, Kendzior M, Nawab A, Caborn DN. Intratunnel versus extratunnel fixation of hamstring autograft for anterior cruciate ligament reconstruction. Arthroscopy. 2012 Oct;28(10):1555-66. doi: 10.1016/j.arthro.2012.02.021. Epub 2012 May 4. PMID 22560484
- [Background] Ilahi OA, Nolla JM, Ho DM. Intra-tunnel fixation versus extra-tunnel fixation of hamstring anterior cruciate ligament reconstruction: a meta-analysis. J Knee Surg. 2009 Apr;22(2):120-9. doi: 10.1055/s-0030-1247736. PMID 19476176
- [Background] Brand J Jr, Weiler A, Caborn DN, Brown CH Jr, Johnson DL. Graft fixation in cruciate ligament reconstruction. Am J Sports Med. 2000 Sep-Oct;28(5):761-74. doi: 10.1177/03635465000280052501. PMID 11032238
- [Background] Hapa O, Barber FA. ACL fixation devices. Sports Med Arthrosc Rev. 2009 Dec;17(4):217-23. doi: 10.1097/JSA.0b013e3181bf668c. PMID 19910779
- [Background] Anderson MJ, Browning WM 3rd, Urband CE, Kluczynski MA, Bisson LJ. A Systematic Summary of Systematic Reviews on the Topic of the Anterior Cruciate Ligament. Orthop J Sports Med. 2016 Mar 15;4(3):2325967116634074. doi: 10.1177/2325967116634074. eCollection 2016 Mar. PMID 27047983
- [Background] Rahr-Wagner L, Lind M. The Danish Knee Ligament Reconstruction Registry. Clin Epidemiol. 2016 Oct 25;8:531-535. doi: 10.2147/CLEP.S100670. eCollection 2016. PMID 27843343
- [Background] Filbay SR, Grindem H. Evidence-based recommendations for the management of anterior cruciate ligament (ACL) rupture. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):33-47. doi: 10.1016/j.berh.2019.01.018. Epub 2019 Feb 21. PMID 31431274
- Available data/document: results can be obtained from principal investigator — https://www.kh-schwaz.at/ — results can be obtained from the principle investigator